CLINICAL TRIAL: NCT06944197
Title: Effectiveness of a Therapeutic Exercise Program of Physiotherapy Through the Use of Telerehabilitation on Functional Capacity for Patients With Chronic Phase Stroke: Multicenter Randomized Controlled Clinical Trial.
Brief Title: Therapeutic Exercise Program of Physiotherapy Using Telerehabilitation on Chronic Phase Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Yaiza Casas, MSc, Physiotherapist, Institut Catala de Salut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/190-P
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Chronic disease; Primary Care; Therapeutic exercises; Telerehabilitation
MeSH Terms: conditions — Stroke; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind study. The research staff who carry out the evaluations will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guiding Document Group (Placebo Comparator): Participating subjects receive a stroke management guide document, as well as guidelines for the promotion and prevention of health of importance after a stroke.
  Interventions: Other: Standard Care Guidance Group
- Therapeutic Exercises Document Group (Active Comparator): The document "Document Therapeutic Exercise Program for the home" will be explained and delivered, which contains an exercise program to be carried out during the next 10 weeks, with a frequency of 3 times a week.
  Interventions: Other: Home-Based Therapeutic Exercise - Document Group
- Telerehabilitation Group (Experimental): An individualized program of therapeutic exercises will be carried out through a Telerehabilitation platform (Physitrack) during the next 10 weeks, with a frequency of 3 times a week.
  Interventions: Other: Home-Based Therapeutic Exercise - Telerehabilitation Group

INTERVENTIONS:
Other: Standard Care Guidance Group — Participants in this group will receive an individual, face-to-face consultation with a physiotherapist from the primary and community care service at the Primary Care Center. During the session, participants will be provided with an informational guide focused on the management of post-stroke conditions, as well as health promotion and secondary prevention strategies relevant to stroke recovery.
  The document provided is titled "Guide for People Affected by Cerebrovascular Disease, Their Families, and Caregivers", published in 2022 by the Department of Health of the Generalitat de Catalunya in collaboration with the Stroke Foundation. This group serves as the control group, as the intervention closely resembles the standard care currently implemented across Primary Care Centers in Catalonia for individuals in the chronic phase of stroke recovery.
  Arms: Guiding Document Group
Other: Home-Based Therapeutic Exercise - Document Group — Participants in this group will receive an individual, face-to-face consultation with a physiotherapist at the Primary Care Center. During the session, the "Home-Based Therapeutic Exercise Program" document will be explained and provided. This document outlines an exercise program to be followed over a 10-week period, with a frequency of three sessions per week.
  The explanatory document includes three weekly exercise charts covering a total of 30 sessions. Each session is clearly described with detailed instructions to ensure proper execution, including dosage specifications such as repetitions, sets, and load. A checklist template is also included to help participants track their progress and completed activities.
  The exercise program consists of strength exercises targeting the major muscle groups of the lower extremities (LE), upper extremities (UE), and trunk; stretching exercises focused on the most relevant flexor muscles of the lower and upper extremities; and exercises aimed
  Arms: Therapeutic Exercises Document Group
Other: Home-Based Therapeutic Exercise - Telerehabilitation Group — Participants will have an individual consultation with a physiotherapist at the Primary Care Center, where an individualized therapeutic exercise program will be explained. The program spans 10 weeks with three sessions per week (totaling 30 sessions) and is delivered through the Physitrack telerehabilitation platform.
  They will receive the "Guide for the Use of the Physitrack Telerehabilitation Platform", which provides all necessary information for effective platform use. A brief tutorial will be given during the consultation to ensure familiarity with the tool.
  The program mirrors the Therapeutic Exercise Document Group program, but with weekly progress monitoring via the platform. This allows the physiotherapist to adjust exercises or load based on progress. The platform also enables direct communication between participants and the physiotherapist, offering continuous support throughout the intervention.
  Arms: Telerehabilitation Group

SUMMARY:
Stroke is the main cause of physical disability in adults in Catalonia. Despite this, there is a lack of evidence on physiotherapy interventions during the chronic phase of the pathology. The objective of the study is evaluate the effectiveness of a therapeutic exercise program of Physiotherapy through the use of Telerehabilitation on functional capacity in activities of daily living in patients with stroke in chronic phase. For this purpose, the investigator conduct a multicenter randomized controlled clinical trial. A minimum of 75 participants will be recruited in three intervention groups (n=25 each group) from Primary Care Centers of the Institut Català de la Salut. The sample will be made up of people over 18 years of age with a medical diagnosis of Stroke, in a chronic phase and with physical sequelae. Research team will evaluate as the main variable the functional capacity for the management of activities of daily living (Barthel Index); as well as sociodemographic variables. Also secondary variables such as motor function (MMAS), muscle tone of affected limbs (MAS), muscle strength of affected limbs (MRC), balance (PASS), gait efficiency (WGS, 4MWT), perception of musculoskeletal pain (BPI), perception of fatigue (FSS), risk of falls (TUG), perception of quality of life (NEWSQOL), and perception of quality of life (NEWSQOL), and perception of perceived subjective change after treatment (GROC). The variables will be collected, before and after the intervention , which will consist of 30 sessions (3 sessions/10 weeks). The analysis will be using a mixed linear model (ANOVA 3X3). Significance level p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Medical diagnosis of stroke
* Stroke condition present for more than 6 months
* Physical sequelae secondary to stroke
* Minimum score of 1 on the Medical Research Council scale for overall muscle strength of affected limbs
* Maximum score of 3 on the Modified Ashworth scale for overall muscle tone of affected limbs
* Maximum score of 4 on the Modified Rankin scale for disability
* Access to computer equipment (tablet, desktop or laptop computer, or smartphone)

Exclusion Criteria:

* Undergoing other non-pharmacological physical treatments for stroke sequelae improvement and/or maintenance
* Previous decreased motor functional capacity with a Barthel scale score of less than 60 points
* Cognitive and/or language barriers that hinder the understanding of informed consent and intervention
* Participation in another clinical trial during the study period that may impact the results of the variables to be evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Level of dependence or functional capacity in activities of daily living (ADLs) | From recruitment to the end of treatment at 10 weeks.
  The primary variable is the degree of dependence or functional capacity in activities of daily living (ADLs), which is assessed using the Barthel Index . This validated scale was also used for sample size calculation. The Barthel Index is a simple, reliable, and valid tool that can detect changes in functional status and is easy to interpret. Despite some limitations, it is widely recommended as a preferred measure for assessing physical disability, both in clinical practice and in epidemiological research and public health. The scale ranges from 0 to 100, where a score of 100 represents complete independence, meaning the person can perform all daily activities without assistance. On the other hand, a score of 0 indicates complete dependence, meaning the person requires full help with these activities. Essentially, higher scores on the Barthel Index reflect better functional independence.

SECONDARY OUTCOMES:
Upper and lower limb motor function | From recruitment to the end of treatment at 10 weeks.
  The Modified Motor Assessment Scale measures motor function in stroke patients, with a particular focus on limb and trunk mobility. This tool evaluates the patient's ability to perform specific motor movements and basic motor activities, providing a measure of motor dysfunction severity and rehabilitation progress. The scale ranges from 0 to 48, where a score of 48 indicates the highest level of motor function, meaning the individual is fully capable of performing the assessed movements independently. A score of 0 indicates the complete inability to perform any of the movements. Higher scores on the MMAS signify better motor function and greater ability to perform voluntary movements."
Upper and lower limb muscle tone | From recruitment to the end of treatment at 10 weeks.
  The Modified Ashworth Scale (MAS) is a widely used and validated tool for assessing muscle tone in stroke patients, particularly to measure the presence and severity of spasticity-an abnormal increase in muscle tone. This scale is specifically designed to evaluate spasticity in patients with neurological impairments, making it highly relevant for stroke rehabilitation.
  The MAS measures the resistance of a muscle to passive movement, providing a score that reflects the degree of spasticity in the patient. The scale ranges from 0 to 4, where 0 indicates no spasticity, and 4 represents extreme rigidity, making it an effective measure for varying levels of spasticity. This tool is particularly useful for assessing patients with moderate to severe spasticity, allowing clinicians to monitor changes over time.
  The interobserver and test-retest reliability of the MAS is generally good, although its subjectivity-since it involves clinical judgment-can lead to variability in results. Despite
Upper amb lower limb muscle strength | From recruitment to the end of treatment at 10 weeks.
  The Medical Research Council (MRC) Scale is a widely utilized tool for assessing muscle strength in patients with various neurological conditions, including stroke. The scale classifies muscle strength on a range from 0 to 5, where 0 indicates the absence of muscle contraction, and 5 represents normal muscle strength with the ability to overcome full resistance against gravity. The MRC Scale demonstrates good interobserver and test-retest reliability, along with strong construct and concurrent validity, making it a robust and effective measure for evaluating muscle function in clinical practice.
Postural Balance | From recruitment to the end of treatment at 10 weeks.
  The Postural Assessment Scale for Stroke Patients (PASS) is a widely used tool designed to assess posture and postural balance in individuals recovering from stroke. It focuses on the patient's ability to maintain and control various postures, which is crucial for motor function recovery during stroke rehabilitation. The scale demonstrates high interobserver and test-retest reliability, as well as strong construct and concurrent validity, correlating well with other established measures of balance and motor function. Additionally, the PASS shows robust predictive validity, effectively identifying patients at higher risk for long-term complications related to balance impairments. The scale ranges from 0 to 36, with higher scores indicating better postural control. A score of 36 suggests the person has normal or near-normal postural stability, meaning they can maintain various positions and perform tasks with minimal difficulty. A score of 0 indicates severe postural instability.
Walking speed and gait performance | From recruitment to the end of treatment at 10 weeks.
  The 4-Meter Gait Speed Test is a straightforward and efficient assessment used to measure a patient's walking speed. Walking speed is closely linked to a variety of functional outcomes, including mobility, independence, and fall risk. This test is known for its high reliability and validity, making it particularly valuable for evaluating gait performance and functional prognosis in stroke patients.
  A faster time (completing the test in fewer seconds) indicates better walking speed and mobility, which are associated with greater functional independence. A slower time may suggest impaired walking ability, which could indicate the need for further rehabilitation or support. Generally, a time of 4 seconds or less is considered normal, while longer times could signal a higher risk of falls or mobility challenges.
Gait performance | From recruitment to the end of treatment at 10 weeks.
  The Wisconsin Gait Scale (WGS) is a tool used to assess aspects of gait, such as postural control, stride length, gait symmetry, and ease of walking. It has high interobserver and test-retest reliability, with good concurrent and predictive validity related to gait, postural control, and fall risk.
  The total score ranges from 0 to 48, with higher scores indicating better gait quality and lower scores indicating more significant gait impairments.
Musculoskeletal pain perception | From recruitment to the end of treatment at 10 weeks.
  The Brief Pain Inventory (BPI) is a widely used tool for assessing both pain intensity and the impact of pain on patients' quality of life. Although initially designed for evaluating pain in cancer patients, its application has expanded to a variety of neurological conditions, including stroke. The BPI is a valid and reliable instrument for measuring pain intensity and its effects on stroke patients. It demonstrates high interobserver and test-retest reliability, enhancing its utility in clinical settings. Furthermore, its construct validity, concurrent validity, and predictive validity affirm its effectiveness in understanding chronic pain and its influence on function and quality of life in stroke patients.
Fatigue perception | From recruitment to the end of treatment at 10 weeks.
  The Fatigue Severity Scale (FSS) is a tool designed to assess the severity of fatigue and its impact on a patient's daily functioning and quality of life. Fatigue is a common and debilitating symptom in stroke patients, significantly affecting their functional capacity and rehabilitation progress. As such, the FSS is widely used to evaluate and monitor this symptom. The scale demonstrates high interobserver and test-retest reliability, making it a valuable tool for both clinical assessment and tracking chronic fatigue in patients. Additionally, its construct validity, concurrent validity, and predictive validity further establish it as an effective measure of the impact of fatigue on stroke patients' quality of life and functional outcomes.
  The Fatigue Severity Scale (FSS) consists of 9 items scored from 1 to 7, with higher scores indicating more severe fatigue. A higher total score, calculated by averaging responses, reflects greater fatigue and its impact on daily life. An FSS score
Fall risk | From recruitment to the end of treatment at 10 weeks.
  The Time Up and Go Test (TUG) is a simple yet effective functional assessment used to evaluate fall risk in patients with various neurological conditions, including stroke. This test measures the time it takes for a patient to stand up from a seated position, walk 3 meters, turn around, return to the chair, and sit down again. The TUG is known for its high interobserver and test-retest reliability, as well as its strong construct, concurrent, and predictive validity, making it an essential tool for both clinical assessment and monitoring progress in post-stroke patients.
  A longer time indicates poorer mobility and higher risk of falls. Typically, a time of 10 seconds or more suggests mobility issues, while times under 10 seconds are considered normal.
Quality of life perception | From recruitment to the end of treatment at 10 weeks.
  The Newcastle Stroke-Specific Quality of Life Measure (NEWSQOL) is a comprehensive assessment tool designed to evaluate stroke-specific quality of life. It captures the impact of stroke on various aspects of a patient's life, including physical, emotional, social, and cognitive dimensions. The tool has been translated into several languages, including Spanish, to ensure broader accessibility. It is a reliable and valid instrument for assessing patients' perception of their quality of life post-stroke. The NEWSQOL demonstrates high internal reliability and test-retest reliability, while its construct validity, concurrent validity, and predictive validity make it an excellent choice for measuring the multifaceted effects of stroke on daily living.
  The Newcastle Stroke-Specific Quality of Life Measure (NEWSQOL) uses a Likert scale (1 to 5) across 12 subscales, with higher scores indicating better quality of life and lower scores reflecting more difficulties following a stroke.
Perception of subjective change post-treatment | From recruitment to the end of treatment at 10 weeks.
  The Global Rating of Change Scale (GROC) is a tool used to assess patients' subjective perception of changes in their health or functioning following an intervention or treatment. In the context of stroke, it measures the perceived improvement or deterioration of a patient's physical, emotional, and functional condition after treatment or rehabilitation. The GROC demonstrates strong test-retest reliability, as well as excellent concurrent and construct validity, making it a valuable tool in both clinical practice and research studies.
  It typically uses a scale from -7 (a very great worsening) to +7 (a very great improvement), with 0 indicating no change. Higher positive scores indicate improvement, while negative scores reflect deterioration.

IPD SHARING:
Plan to Share IPD: No